CLINICAL TRIAL: NCT06599229
Title: Myocardial Perfusion Abnormalities in Hypertrophic Cardiomyopathy
Brief Title: Perfusion Abnormalities in Hypertrophic Cardiomyopathy
Status: Not yet recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jonathan Lindner, MD, Professor of Medicine, University of Virginia
Other Study IDs: 301910
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: hypertrophic cardiomyopathy; myocardial contrast echocardiography; microvascular perfusion
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HCM initiated on cardiac myosin inhibitor therapy: Patients with HCM who are being initiated on cardiac myosin inhibitor therapy for clinically indicated reasons.
  Interventions: Diagnostic Test: myocardial contrast echo

INTERVENTIONS:
Diagnostic Test: myocardial contrast echo — Vasodilator stress myocardial contrast echocardiography will be performed at baseline and within 4 months of reaching target dose of a cardiac myosin inhibitor.

SUMMARY:
The purpose of this study is to investigate whether myocardial microvascular perfusion in patients with hypertrophic cardiomyopathy improved after initiation of cardiac myosin inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertrophic cardiomyopathy
* Subject being initiated on clinically-indicated cardiac myosin inhibitor therapy

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy to ultrasound enhancing agent (lipid-stabilized) or regadenoson
* Serious AE to regadenoson
* Hypotension
* Serious bradycardia not addressed by pacemaker
* Moderate or greater reactive airways disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCM who are being started on cardiac myosin inhibitor therapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Peak hyperemic perfusion | 3 months
  Myocardial contrast echo-derived myocardial blood flow at peak hyperemia (produced by regadenoson)

SECONDARY OUTCOMES:
Resting myocardial perfusion | 3 months
  Resting myocardial perfusion by MCE

IPD SHARING:
Plan to Share IPD: Yes
De-identified data on patient demographics, HCM type, medication dose, transthoracic echo data, MCE perfusion imaging data at rest and during regadenoson
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2024; End-date not determined but no sooner than December 2028
Access Criteria: Any investigators requesting access to data after publication of results.